CLINICAL TRIAL: NCT05837819
Title: Methodology Issues in a Tailored Light Treatment for Persons With Dementia - Aim 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Mariana Figueiro, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-20-01736 Aim 2
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer's Disease; Sleep Disturbance
MeSH Terms: conditions — Alzheimer Disease; Parasomnias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Lighting Intervention (Active Comparator): Lighting intervention designed to effect the circadian system then will receive the control lighting intervention.
  Interventions: Device: Active Lighting Intervention; Device: Control Lighting Intervention
- Control Lighting Intervention (Placebo Comparator): Lighting intervention using low light levels designed to not effect the circadian system
  Interventions: Device: Control Lighting Intervention

INTERVENTIONS:
Device: Active Lighting Intervention — Lighting intervention using high light levels designed to effect the circadian system
  Arms: Active Lighting Intervention
Device: Control Lighting Intervention — Lighting intervention using low light levels designed to not effect the circadian system

SUMMARY:
Aim 2 will investigate the effect of 3 different light exposure lengths on sleep, mood and agitation in persons with Alzheimer's disease. Participants will be randomly assigned to one of three conditions of light exposure: 1) 2-h morning light exposure; 2) 4-h morning light exposure; and 3) all day light exposure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's disease or related dementia with a Montreal Cognitive Assessment score <25
* Sleep disturbance with a Pittsburgh Sleep Quality Index score ≥5

Exclusion Criteria:

* Extensive brain vascular disease, traumatic brain injury, multiple sclerosis, Parkinson's Disease
* Obstructing cataracts
* Severe macular degeneration
* Use of sleep medication
* Use of oral melatonin
* untreated moderate to severe sleep apnea
* Severe restless leg syndrome
* Blindness

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 135 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Sleep Disturbance using the Pittsburgh Sleep Quality Index | up to week 14
  The PSQI is used to measure sleep quality and is composed of 19 items that generate 7 component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction). Each subscale is scored 0 to 3. The sum of the 7 component scores yields a single global score with a range of 0 to 21. A higher score indicates higher sleep disturbance

SECONDARY OUTCOMES:
Sleep efficiency using actigraphy | up to week 14
  Actigraphs will be worn continuously for 7 days during each assessment week. Changes in sleep efficiency will be measured using the actigraphy software. Sleep efficiency is a calculated as a ratio of the time spent in bed and the time spent sleeping.
Depression using the Cornell Scale for Depression in Dementia (CSDD) | up to week 14
  The CSDD is a 19-item tool designed to rate symptoms of depression in patients with dementia. This tool evaluates the presence and extent of mood-related signs (anxiety, sadness, irritability), behavioral disturbances (agitation, loss of interest), physical signs (loss of appetite, weight loss), cyclic functions (mood variation, sleep quality), and ideational disturbances. Scores range from 0 to 38 with a higher score indicating greater depression.
Agitation using the Cohen-Mansfield Agitation Inventory (CMAI) | up to week 14
  The CMAI assesses the frequency of manifestations of agitated behaviors in elderly persons. The CMAI is a caregivers' rating questionnaire consisting of 29 agitated behaviors, each rated on a 7-point scale of frequency. Score ranges from 30 to 210 with a higher score indicating higher agitated behavior.
Light measurements using the Daysimeter | up to week 14
  Circadian light measurements will be collected during waking hours for 7 days each assessment week using the daysimeter. The light measurement is reported as Lux levels.
Cognitive status Using the Montreal Cognitive Assessment (MOCA) | up to week 14
  The MoCA is a 1-page, 30-point test that can be administered in 10 minutes. It assesses short-term memory, visuospatial abilities, executive functions, attention, concentration and working memory, language, and orientation to time and place. Total score range from 0 to 30. Lower score indicates lower cognitive status.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Figueiro, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, Albany, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No
Overall results will be shared, not individual data